CLINICAL TRIAL: NCT02689869
Title: A Chemotherapy-free Combination of the Bruton's Tyrosine Kinase Inhibitor, Ibrutinib in Combination With GA 101 in Patients With Previously Untreated Follicular Lymphoma and a High Tumor Burden
Brief Title: Combination of PCI-32765 With Obinutuzumab in Untreated Follicular Lymphoma
Acronym: Alternative
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Hoffmann-La Roche (Industry); Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Hiddemann, Prof. Dr. med. W. Hiddemann, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-005164-15
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Indolent Non-Hodgkin Lymphoma
Keywords: indolent lymphoma; novel agents; chemotherapy free treatment; ibrutinib; obinutuzumab; GA101
MeSH Terms: interventions — ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib and GA 101 (Experimental): Initial therapy 6 cycles of Ibrutinib:
  Ibrutinib 560 mg once daily every day until start of maintenance for a total of 24 weeks.
  1000 mg of GA101 I.V. on days d 1, 8, 15 of cycle 1 and on day 1 of cycles 2-6 (21 day cycles).
  Maintenance with another 24 months of ibrutinib plus GA101 in patients with clinical remission after the last induction cycle:
  Ibrutinib 560 mg once daily every day. GA101 at a dose of 1000 mg I.V. every 2 months for a total of 24 months. The total duration of ibrutinib plus obinutuzumab therapy will therefore be 30 months.
  In patients remaining MRD positive at 30 months without clinical progression, single agent ibrutinib therapy is continued for another 12 months.
  Interventions: Drug: Ibrutinib; Drug: GA 101

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib (PCI-32765; JNJ-54179060) is a first-in-class, potent, orally-administered covalently-binding small molecule inhibitor of Bruton's tyrosine kinase currently being co-developed by Janssen Research & Development, LLC and Pharmacyclics, Inc for the treatment of B-cell malignancies.
  Other Names: Imbruvica
Drug: GA 101 — Obinutuzumab (GA 101) is a first-in-class, potent, intravenously administered type II anti-CD 20 antibody that is developed by Roche AG for the treatment of B-cell malignancies.
  Other Names: Obinutuzumab

SUMMARY:
Primary Objectives The primary objective of this study is to evaluate the efficacy of the chemotherapy-free combination of ibrutinib and obinutuzumab (GA 101) in patients with previously untreated follicular lymphoma (FL) and a high tumor burden. Primary endpoint to be observed for this is the rate of progression free survival one year after start of therapy.

Hypothesis The hypothesis of the study is that ibrutinib in combination with obinutuzumab will achieve response rates (CR and PR), rates of MRD negativity and PFS which are comparable to currently used standard rituximab-chemotherapy combinations such as R-CHOP or R-bendamustine in subjects with previously untreated FL and a high tumor burden.

DETAILED DESCRIPTION:
OVERVIEW OF STUDY DESIGN This is a prospective, multicenter phase 2 study in up to 98 subjects with previously untreated FL and a high tumor burden in advanced stages and in need of therapy. The study will include a central monitoring of MRD by PCR, a central pathologic review and complimentary research projects including monitoring of immune response.

The study therapy comprises an initial 6 cycles of ibrutinib plus obinutuzumab followed by an additional 24 months of ibrutinib plus obinutuzumab maintenance.

In patients being MRD negative at 30 months, i.e. at the end of ibrutinib plus obinutuzumab maintenance, and without clinical progression no further treatment is given while MRD monitoring is continued.

MRD monitoring will be regularly performed on peripheral blood samples collected before the start of therapy and at months 3, 6, 9, 12, 18, 24 and 30 respectively. Subsequently, MRD analyses will be performed every 6 months until clinical progression of the disease or for a maximum of 4 years (until the end of the study).

If MRD assessment on peripheral blood samples turns from positive to negative within the first 30 months, confirmatory blood and bone marrow samples should be taken 6 months thereafter.

In patients remaining MRD positive at 30 months without clinical progression, single agent ibrutinib therapy is continued for another 12 months.

An independent Data Monitoring Committee (DMC) will be formed and constituted. The independent DMC will review the safety of the treatment and make recommendations as to the further conduct of the study.

The data generated by this phase II study should serve as the basis for a subsequent randomized phase III study comparing the chemotherapy-free combination of ibrutinib plus obinutuzumab with standard immune-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed follicular lymphoma grade 1, 2 or 3A with a lymph node biopsy performed within 12 months before study entry and with material available for central review and complementary scientific analyses

* Ann Arbor stage III/IV, or stage II not suitable for radiotherapy, or stage II bulky disease
* Age ≥ 18 years
* No prior lymphoma therapy
* Need for start of therapy as defined by:

  * bulky disease at study entry according to the GELF criteria (nodal or extranodal mass >7 cm in its greater diameter)
  * and/or B symptoms (fever, drenching night sweats, or unintentional weight loss of >10% of normal body weight over a period of 6 months or less)
  * and/or hematopoietic insufficiency (granulocytopenia < 1.500/µl, Hb < 10 g/dl, thrombocytopenia < 100.000/µl)
  * compressive syndrome or high risk for compression syndrome
  * and/or pleural/peritoneal effusion
  * and/or symptomatic extranodal manifestations
* At least one bi-dimensionally measurable lesion (> 2 cm in its largest dimension by CT scan or MRI)
* Performance status ≤ 2 on the ECOG scale
* Adequate hematologic function (unless abnormalities are related to NHL), defined as follows:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1500 /µl
  * Platelet count ≥ 75000 /µl
* Women are not breast feeding, are using highly effective contraception, are not pregnant, and agree not to become pregnant during participation in the trial and during the 18 months thereafter (pregnancy testing is mandatory for premenopausal women).
* Men agree not to father a child during participation in the trial and during the 18 months thereafter.
* Written informed consent

Exclusion Criteria:

* - Transformation to high-grade lymphoma (secondary to "low grade" FL)
* Grade 3B follicular lymphoma
* Presence or history of CNS disease (either CNS lymphoma or leptomeningeal lymphoma).
* Known hypersensitivity to any of the study drugs
* Known sensitivity to murine products
* Regular use of corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 20 mg/day prednisone.
* Concomitant use of strong CYP3A4 inhibitors and / or oral anticoagulants (warfarin and/or phenprocoumon)
* Prior or concomitant malignancies except:

  * non-melanoma skin cancer or adequately treated in carcinoma in situ of the cervix
  * Other malignant diseases not specified above which have been curatively treated by surgery alone and from which subject is disease-free for ≥5 years without further treatment
* Serious disease interfering with a regular therapy according to the study protocol:

  * Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
  * pulmonary (e.g. chronic lung disease with hypoxemia)
  * endocrine (e.g. severe, not sufficiently controlled diabetes mellitus)
  * renal insufficiency (unless caused by the lymphoma): creatinine > 2x normal value and/or creatinine clearance < 50 ml/min)
  * impairment of liver function (unless caused by the lymphoma): transaminases > 3x normal or bilirubin > 2,0 mg/dl (unless caused by known Morbus Meulengracht [Gilbert-Meulengracht-Syndrome])
* Positive test results for chronic HBV infection (defined as positive HBsAg serology) Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible.
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing). Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Known history of HIV seropositive status.
* Patients with a history of confirmed PML
* Vaccination with a live vaccine within 28 days prior to registration
* Recent major surgery (within 4 weeks prior to the start of Cycle 1)
* History of stroke or intracranial hemorrhage within 6 months prior to registration
* Serious underlying medical conditions, which could impair the ability of the patient to undergo the treatment offered in the study (e.g. ongoing infection, gastric ulcers, active autoimmune disease)
* Treatment within a clinical trial within 30 days prior to trial entry.
* Prior organ, bone marrow or peripheral blood stem cell transplantation
* Known or persistent abuse of medication, drugs or alcohol
* Any other co-existing medical or psychological condition that will preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-04; Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | one year progress free survival
  The rate of patients archiving a progression free survival of more than one year after registration (one-year PFS) will serve as early readout for efficacy and will be the primary endpoint of this trial.

SECONDARY OUTCOMES:
three-year-PFS | three years after start of therapy
  Progression free survival after start of therapy (continuous observation)
  * three-year-PFS
CR | one year after start of therapy and at 30 months after end of maintenance
  CR rates at end of induction CR rates one year after start of therapy CR rates after end of maintenance therapy (at 30 months after start of therapy: CR30)
PR | one year after start of therapy and at 30 months after end of maintenance
  PR rates at end of induction PR rates one year after start of therapy PR rates after end of maintenance therapy (at 30 months after start of therapy: CR30)
SD | one year after start of therapy and at 30 months after end of maintenance
  SD rates at end of induction
Duration of response | 4,5 up to 6,5 years through study completion
  Duration of Response
Percentage of Progression | 4,5 up to 6,5 years through study completion
  Percentage of progression during induction and maintenance therapy
TTF after start of therapy | 4,5 up to 6,5 years through study completion
  Time to treatment failure after start of therapy (failure defined by failure to achieve a CR/PR after 6 months or progression after CR or PR or death in remission)
Time to next anti-lymphoma therapy / time to next chemotherapy based treatment | 4,5 up to 6,5 years through study completion
  Time to next anti-lymphoma therapy and time to next chemotherapy based treatment
Treatment associated adverse events | 4,5 up to 6,5 years through study completion
  Treatment associated adverse events
Percentage of MRD negative patients during therapy | 4,5 up to 6,5 years through study completion
  Percentage of MRD negative patients during induction therapy (midterm), after induction therapy and after maintenance therapy
Duration of molecular remission | 4,5 up to 6,5 years through study completion
  Duration of molecular remission for MRD negative patients after the end of induction and maintenance
Percentage of secondary transformation | 4,5 up to 6,5 years through study completion
  Percentage of secondary Transformation to aggressive lymphoma
Percentage of secondary malignancies | 4,5 up to 6,5 years through study completion
  Percentage of secondary malignancies
Time to first secondary malignancy | 4,5 up to 6,5 years through study completion
  Time to first secondary malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hiddemann, Prof., Principal Investigator — Klinikum der Universität München
Locations (1):
- Klinikum der Universität München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No